CLINICAL TRIAL: NCT01870258
Title: Prediction of Acute Myocardial Infarction With Artificial Neural Networks in Patients With Nondiagnostic Electrocardiogram
Brief Title: Myocardial Infarction Prediction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 90-8037
Record Dates: First submitted 2013-05-24; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Myocardial Infarction; Artificial Neural Network
Keywords: Myocardial infarction; artificial neural networks; Electrocardiography
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- those without MI in 2 weeks (Placebo Comparator): patient without MI in 2 weeks
  Interventions: Other: ANN prediction of myocardial infarction
- patient with MI (Active Comparator): group with MI in 2 weeks
  Interventions: Other: ANN prediction of myocardial infarction

INTERVENTIONS:
Other: ANN prediction of myocardial infarction
  Other Names: sofware detected risk of new myocardial infraction

SUMMARY:
prediction of MI in patients with chest pain and nondiagnostic ECG was done in 2 weeks

DETAILED DESCRIPTION:
Myocardial infarction remains one the leading causes of mortality and morbidity and involves a high cost of care. Early prediction can be helpful in preventing the development of myocardial infarction with appropriate diagnosis and treatment. Artificial neural networks have opened new horizons in learning about the natural history of diseases and predicting cardiac disease.

Methods: A total of 935 cardiac patients with chest pain and nondiagnostic electrocardiogram (ECG) were enrolled and followed for 2 weeks in two groups based on the appearance of myocardial infarction. Two types of data were used for all patients: nominal (clinical data) and quantitative (ECG findings). Two different artificial neural networks - radial basis function (RBF) and multi-layer perceptron (MLP) - were used.

ELIGIBILITY:
Inclusion Criteria:

* patient with chest pain refered to ER with nondiagnostic ECG

Exclusion Criteria:

* 1) Absence of a history of myocardial infarction
* 2) Absence of bundle branch block, Wolf-Parkinson-White abnormality, ventricular hypertrophy or previous ECG signs of myocardial infarction,
* 3) Absence of a history of percutaneous coronary surgery or coronary artery bypass grafting,
* 4) Absence of ECG abnormalities attributable to drugs such as digoxin or tricyclic antidepressants.

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | 2 weeks

SECONDARY OUTCOMES:
hospital admission due to cardiac events | 2 weeks
  may be includes unstable angina, cardiac arrest or PCIor CABG